CLINICAL TRIAL: NCT02856698
Title: Study Design and Rationale of "A Multicenter, Open-Labeled, Randomized Controlled Trial Comparing MIdazolam Versus MOrphine in Acute Pulmonary Edema": MIMO Trial
Brief Title: MIdazolam Versus MOrphine in Acute Pulmonary Edema (MIMO Trial)
Acronym: MIMO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped because of the adverse events
Sponsor: Alberto Dominguez-Rodriguez (Other)
Responsible Party: Sponsor-Investigator, Alberto Dominguez-Rodriguez, Alberto Domínguez- Rodríguez, MD, PhD, FESC, Hospital Universitario de Canarias
Organization: Hospital Universitario de Canarias (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT: 2016-000884-17
Record Dates: First submitted 2016-07-20; First posted 2016-08-05 (Estimated); Results first posted 2022-05-19 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Acute Pulmonary Edema
Keywords: Acute heart failure; morphine; midazolam; in-hospital mortality
MeSH Terms: interventions — Midazolam; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- midazolam (Experimental): The dose of midazolam intravenously will be of 1 mg which may be repeated until a total dose of 3 mg.
  Interventions: Drug: Midazolam
- morphine (Active Comparator): The dose of morphine intravenously is of 2-4 mg which may be repeated until a total dose of 8 mg if the patient continue suffering from severe anxiety or distress caused by APE
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Midazolam — Dose use according to the product technical sheet
  Arms: midazolam
Drug: Morphine — Dose use according to the product technical sheet
  Arms: morphine

SUMMARY:
Acute pulmonary edema (APE) is a common condition in the emergency room, associated with considerable mortality. The use of intravenous morphine in the treatment of APE remains controversial and Benzodiazepines have been suggested as an alternative for morphine to relieving dyspnoea and anxiety in the patients with APE. The MIdazolan versus MOrphine in APE trial (MIMO) is a multicenter, prospective, open-label, randomized study designed to evaluate the efficacy and safety of morphine in patients with APE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pulmonary edema with dyspnoea and anxiety

Exclusion Criteria:

* Patients with known severe liver disease.
* Patients with known severe renal disease.
* Patients with expectation of death from other illness during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-04-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Universitario Reina Sofía de Córdoba, Córdoba, Andalusia
  - Hospital Comarcal de la Axarquía, Málaga, Andalusia
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital General de Alicante, Alicante
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Comarcal de Axarquia, Málaga
  - Hospital General Universitario Reina Sofía, Murcia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period goes from 08/04/2017 to 30/12/2020
Period: Overall Study
Arm/Group | Midazolam | Morphine
Started | 55 | 56
Completed | 48 | 46
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Population: All quantitative and categorical variables were expressed as median (interquartile range) and n (%) and were compared using the Mann-Whitney U test and Fisher's exact test respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Morphine | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Categorical [Count of Participants; unit: Participants] — All quantitative and categorical variables were expressed as median (interquartile range) and n (%) and were compared using the Mann-Whitney U test and Fisher's exact test respectively.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 7 | 16
    >=65 years | 46 | 49 | 95
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 78.4 [67.8 to 83.1] | 79.9 [75.8 to 83.9] | 79.15 [71.8 to 83.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 27 | 26 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 55 | 56 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: In-hospital Mortality
Description: In hospital mortality
Time Frame: 28 days after of the hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Morphine
Number analyzed (Participants) | 55 | 56
Participants | 7 | 10

2. Secondary Outcome: Number of Participants That Required Invasive Mechanical Ventilation
Time Frame: Up to 1 week
Measure: Number; unit: participants
Arm/Group | Midazolam | Morphine
Number analyzed (Participants) | 55 | 56
participants | 3 | 1

3. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Midazolam | Morphine
Number analyzed (Participants) | 55 | 56
days | 7 [5 to 14] | 6 [4 to 13]

ADVERSE EVENTS:
Time Frame: The adverse events were collected through study completion (1 year)
Description: The adverse events observed were related to the circulatory, respiratory, and other systems (nervous, endocrine and renal).
Arm/Group | Midazolam | Morphine
All-Cause Mortality (participants affected / at risk) | 9/55 | 13/56
Serious Adverse Events (participants affected / at risk) | 10/55 | 24/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=55) | Morphine (N=56)
ischemic stroke (Cardiac disorders) | 10 (10) | 24 (24) — Patient with capsular lacunar infarction three days after receiving study treatment for acute lung edema which is the disease under study in the clinical trial

LIMITATIONS AND CAVEATS:
The main limitation of the study was that the study treatment, because it was a serious pathology, was sometimes administered in the ambulance, before admission to the hospital emergency room.

Another limitation has been the COVID-19 pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT02856698/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02856698/SAP_001.pdf